CLINICAL TRIAL: NCT04398381
Title: One-year Outcome of Critically Ill Patients With Systemic Rheumatic Disease: a Multicenter Cohort Study
Brief Title: Prognosis of SRD Patients in the ICU
Acronym: ProSyDICU
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); Sorbonne University (Other); Hôpital Lariboisière Fernand Widal (Other); Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0289
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Systemic Rheumatic Diseases; Intensive Care Unit; Corticosteroids
Keywords: outcomes; prognostic factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critically ill systemic rheumatic disease (SRD) patients have benefited from better provision of rheumatic and critical care in recent years. Recent comprehensive data regarding in-hospital mortality and most importantly long-term outcome are scarce. The aim of this study is to assess short and long-term outcome of patients with SRD admitted to the ICU in a retrospective cohort study (2006 - 2016).

ELIGIBILITY:
Inclusion criteria:

* All consecutive SRD patients admitted to ICUs during the study period
* at least one urine sample

Exclusion criteria:

* Age < 18 years
* Persons under protection
* Paritcipation rejections
* Admition to the ICU after scheduled surgery or trauma or suicide attempt unrelated to neurological involvement of SRD
* Cancer treated with chemotherapy within a month before ICU admission

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive SRD patients admitted to ICUs during the study period
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate in the ICU associated risk factors | 1 day
  Mortality rate in the ICU associated risk factors

SECONDARY OUTCOMES:
Mortality rate in the hospital and one-year after ICU admission and associated risk factors | 1 day
  Mortality rate in the hospital and one-year after ICU admission and associated risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Romaric Larcher, MD PhD, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC